CLINICAL TRIAL: NCT01242579
Title: A Double-Blind, Randomised, Placebo-Controlled Phase I Trial to Compare the Pharmacokinetics of Maraviroc and Dapivirine Following Application of Maraviroc Vaginal Vaginal Gel, 0.1% 2.5g, Dapivirine Vaginal Gel, 0.05%, 2.5g and Maraviroc 0.1% + Dapivirine 0.05% Vaginal Gel, 2.5g Formulations, and to Assess Their Safety as Compared to the Matching Placebo Vaginal Gel, 2.5g in Healthy, HIV-Negative Women
Brief Title: A Safety and Pharmacokinetic Study for Dapivirine and Maraviroc Gel in Belgium
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: In order to focus efforts on the combination ring formulation, IPM decided not to move forward with this trial.
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Annalene Nel, MBChB, PhD, IPM
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 025
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Maraviroc Vaginal Gel (Active Comparator): Drug: Maraviroc dosage form: vaginal gel dosage: 2.5g frequency: once daily duration: 11 days
  Interventions: Drug: Maraviroc Vaginal Gel
- Dapivirine Vaginal Gel (Active Comparator): Drug: Dapivirine dosage form: vaginal gel dosage: 2.5g dapivirine frequency: once daily duration: 11 days
  Interventions: Drug: Dapivirine Vaginal Gel
- Matching Placebo Gel (Placebo Comparator): Drug: placebo dosage form: vaginal gel dosage: 2.5g placebo frequency: once daily duration: 11 days
  Interventions: Drug: Matching Placebo Gel
- Maraviroc/Dapivirine Gel (Experimental): Drug: Maraviroc/Dapivirine dosage form: combination vaginal gel dosage: 2.5g - Maraviroc 0.1%, Dapivirine 0.05% frequency: once daily duration: 11 days
  Interventions: Drug: Maraviroc/Dapivirine Gel

INTERVENTIONS:
Drug: Maraviroc/Dapivirine Gel — Vaginal gel containing 2.5g - Maraviroc 0.1%, Dapivirine 0.05%
  Arms: Maraviroc/Dapivirine Gel
Drug: Dapivirine Vaginal Gel — Dapivirine vaginal gel containing 2.5g
  Arms: Dapivirine Vaginal Gel
Drug: Maraviroc Vaginal Gel — Maraviroc vaginal gel containing 2.5g
  Arms: Maraviroc Vaginal Gel
Drug: Matching Placebo Gel — Matching placebo gel containing 2.5g
  Arms: Matching Placebo Gel

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of the combination dapivirine and maraviroc gel and determine whether it is safe for daily use by healthy women in the United Kingdom

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to40 years of age who can give written informed consent (illiterate participants may provide a thumbprint or mark witnessed and signed by a person independent from trial staff);
* Available for all visits and consent to follow all procedures scheduled for the trial;
* HIV-negative as determined by an HIV test at time of enrollment;
* Be on a stable form of contraception, defined as:
* A stable oral contraceptive regimen for at least 2 months prior to enrollment, OR,
* Transdermal contraceptive patch for at least 3 months prior to enrollment, OR,
* Long-acting progestins for at least 6 months prior to enrollment, OR,
* An IUD inserted (with no vaginal or gynaecological complaints associated with its use) at least 3 months prior to enrolment, OR,
* Have undergone surgical sterilization at least 3 months prior to enrollment;
* In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle, defined as having a minimum of 21 days and a maximum of 35 days between menses;
* Upon pelvic examination and colposcopy at the time of enrollment, the cervix and vagina appear normal as determined by the Investigator;
* Asymptomatic for genital infections at the time of enrollment (if a woman is diagnosed with any treatable STI, either syndromically or by laboratory test at the time of screening, she must receive treatment at least 2 weeks prior to enrollment and have completed treatment);
* Willing to refrain from the use of vaginal products or objects including, tampons, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 14 days prior to enrollment and for the duration of the trial;
* Willing to use oral contraceptives to avoid menstruation, if necessary, while taking part in this trial;
* Documentation of no abnormality on Pap test, including grossly bloody smear, within 3 months prior to screening;
* Willing to refrain from participation in any other research trial for the duration of this trial;
* Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures [e.g., by home visit or telephone; or via family or close neighbour contacts (confidentiality to be maintained)];
* Willing to agree to abstain from oral contact with her genitalia for gel use period, as well as for a total of 3 days (72 hours) after the biopsy procedure:
* Willing to remain sexually abstinent for the gel use period in this trial;
* Hepatitis B and C negative at the time of enrollment.

Exclusion Criteria:

* Currently pregnant or having had their last pregnancy outcome within 3 months prior to screening;
* Currently breast-feeding;
* Currently or within two months of participation in any other clinical research trial involving investigational or marketed products prior to screening;
* Untreated symptomatic urogenital infections, e.g., urinary tract or other sexually transmitted infections, or other gynaecological conditions such as vaginal itching, pain, or discharge, within 2 weeks prior to enrolment;
* Presence of any abnormal clinically significant physical finding on the vulva, vaginal walls or cervix during pelvic examination and/or colposcopy at pre-enrolment;
* History of urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence;
* Current vulvar or vaginal symptoms/abnormalities that could influence the trial results;
* Pap test result that requires cryotherapy, biopsy, treatment (other than for infection); or further evaluation [this includes any findings of atypical squamous cells of undetermined significance (ASCUS)];
* Symptomatic genital HSV infection or a history of genital herpetic infection;
* Any Grade 2, 3 or 4 haematology, chemistry or urinalysis laboratory abnormality at baseline (screening) according to the DAIDS Table for Grading Adverse Events (NOTE: This table can be found at: http://rcc.tech-res.com/safetyandpharmacovigilance;and a standardized version will be provided to the research centre in the Study Operations Manual);
* Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrollment;
* Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone;
* Any serious acute, chronic or progressive disease (e.g., any known history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, HIV, AIDS, or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition;
* Have undergone a hysterectomy;
* History of drug abuse within 1 year of enrollment;
* Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety: To assess the safety and tolerability of the combination maraviroc and dapivirine gel, the endpoint was the proportion of women in the four arms experiencing specific, protocol defined safety events during the study (see description). | 8 weeks
  * Mucosal abnormalities (as defined in the WHO/CONRAD manual) visible during naked eye examination and/or colposcopy;
  * Abnormal vaginal pH and/or abnormal vaginal flora during the course of the trial;
  * Positive diagnostic tests for trichomonas, gonorrhoea and/or chlamydia;
  * At least one adverse event during the 2 month trial period;
  * Any laboratory abnormalities on haematology, electrolytes, liver function, and renal function.
Pharmacokinetics: assessment of local and systemic pharmacokinetics of maraviroc and dapivirine in plasma, vaginal fluid and cervical tissue before, during and after 11 days. | 8 weeks